CLINICAL TRIAL: NCT00396916
Title: The Value of Novel Imaging Modality, Hybrid PET/CT, Using F18-Flurodeoxyglucose(FDG) in the Assessment of Cancer Patients. Impact of PET/CT on Clinical Management of Patients With Rising Tumor Markers and no Other Evidence of Disease and in Patients With Metastatic Cancer of Unknown Origin
Brief Title: Hybrid PET/CT in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: hybridCTIL
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-04

CONDITIONS: Cancer
Keywords: cancer patients
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Device: PET/CT imaging

SUMMARY:
The purpose of the present study is to assess the role of hybrid PET/CT imaging diagnosis of active malignancy in cancer patients with rising tumor markers after treatment and in the diagnosis of primary tumor in patients with metastatic cancer of unknown origin. The clinical impact of PET/CT in the management and treatment of these two groups of cancer patients will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients in complete remission after treatment, with serial elevation of serum tumor markers and negative CT or other conventional imaging test.
* Patients with newly diagnosed metastatic cancer with unknown primary tumor
* Glucose levels below 150-200
* Patient signed informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Patient unable or not willing to tolerate the test until its completion
* One or more of the inclusion criteria is not fulfilled

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45
Dates: Start 2004-12

PRIMARY OUTCOMES:
the impact of the imaging modality on patient management

SECONDARY OUTCOMES:
the impact of the imaging modality on patient management

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Bar-Shalom, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel